CLINICAL TRIAL: NCT01923792
Title: An Optional Follow-Up Study to Evaluate the Continued Efficacy of ToleroMune HDM in House Dust Mite Allergic Subjects Following Challenge With House Dust Mite Allergen in an Environmental Exposure Chamber
Brief Title: ToleroMune House Dust Mite Follow on Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Inflamax Research Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: TH002a
Record Dates: First submitted 2013-07-16; First posted 2013-08-16 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: House Dust Mite Allergy; Rhinoconjunctivitis
Keywords: House Dust Mite Allergy; Rhinoconjunctivitis; Environmental Exposure Unit; Immunotherapy; ToleroMune HDM
MeSH Terms: conditions — Dust Mite Allergy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Placebo: Subjects previously randomised to receive placebo in study TH002
- ToleroMune HMD Group 1: Subjects previously randomised to receive ToleroMune HDM in study TH002
- ToleroMune HDM Group 2: Subjects previously randomised to receive ToleroMune HDM in study TH002

SUMMARY:
House Dust Mites (HDM) are arachnids that infest bedding, carpet, upholstered furniture and fabric. Like many other allergens, exposure to HDM allergens in sensitised patients is associated with poorer lung function, greater medication requirements and more asthma symptoms as well as chronic rhinosinusitis symptoms. In contrast to other allergens, there is evidence that HDMA leads to the development of asthma, in addition to exacerbating pre-existing asthma in HDM-sensitised patients.

ToleroMune HDM is currently being developed for the treatment of HDM allergy.

The Purpose of this optional observational follow-on study is to evaluate the continued efficacy of TM-HDM in HDM allergic subjects based on change in TRSS from TH002 baseline approximately two years after the completion of the baseline EEC visit in TH002 following challenge with HDM allergen in an EEC.

DETAILED DESCRIPTION:
Subjects who completed all dosing visits and the post treatment challenge (PTC) in study TH002 will be invited to attend the Screening visit for TH002a. Subjects will attend for 3 visits to the EEU on successive days. Following the last EEC visit a follow-up visit will be performed 3-10 days later.

ELIGIBILITY:
Inclusion Criteria:

* previously randomised in study TH002, completed all dosing visits and the PTC

Exclusion Criteria:

* "Partly controlled" and "uncontrolled" asthma
* History of anaphylaxis to House Dust Mite allergen
* FEV1 <80% of predicted.
* Symptoms of a clinically relevant illness
* Subjects who cannot tolerate allergen challenge in the EEC

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects previously randomised in study TH002 and completed all dosing visits and the PTC
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Scores | 2 years post after the completion of the baseline environmental exposure chamber (EEC) visit in TH002

SECONDARY OUTCOMES:
Total Nasal Symptom Scores (TNSS) | Two years after the completion of the baseline EEC visit in TH002
Der p Specific IgA | Two years after the completion of the baseline EEC visit in TH002
Total Non Nasal Symptom Scores (TNNSS) | Two years after the completion of the baseline EEC visit in TH002
Der P Specific IgE | Two years after the completion of the baseline EEC visit in TH002
Der p specific IgG4 | Two years after the completion of the baseline EEC visit in TH002